CLINICAL TRIAL: NCT00254839
Title: Bacterial Accumulation and Malodor Production in Various Types of Dental Implants
Brief Title: Association Between Dental Implants Properties and Malodor Production
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: 01-05-HMO-CTIL
Record Dates: First submitted 2005-11-16; First posted 2005-11-17 (Estimated); Last update posted 2006-09-15 (Estimated); Status verified 2005-11

CONDITIONS: Halitosis
Keywords: Oral malodor; Dental implants
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Malodor production is bacterial in origin. The bacterial activity of anaerobic bacteria results in the breakdown of proteins and the production of foul smelling compounds. The aim of the study is to test the hypothesis that bacterial growth on dental implants contributes to malodor production and to see whether this contribution is associated with various properties of the dental implant such as: maker, type, depth ext.

ELIGIBILITY:
Inclusion Criteria:Dental patients that need dental implants -

Exclusion Criteria:smokers

-

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Nir Sterer, Dr., Principal Investigator — Hadassah - Hebrew University School of Dental medicine
Locations (1):
- Hadasssah Medical Organization, Jerusalem, Israel